CLINICAL TRIAL: NCT02247479
Title: A Phase III, Multicenter, Randomized, Double-Masked, Sham-Controlled Study to Assess the Efficacy and Safety of Lampalizumab Administered Intravitreally to Patients With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Brief Title: A Study Investigating the Efficacy and Safety of Lampalizumab Intravitreal Injections in Participants With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Acronym: CHROMA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GX29176; 2014-000107-27 (EudraCT Number)
Record Dates: First submitted 2014-07-15; First posted 2014-09-25 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy | interventions — lampalizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lampalizumab Once in Every 4 Weeks (Q4W) (Experimental): Participants will receive 10 milligrams (mg) dose of lampalizumab administered by intravitreal injections for approximately 96 weeks.
  Interventions: Drug: Lampalizumab
- Lampalizumab Once in Every 6 Weeks (Q6W) (Experimental): Participants will receive 10 mg dose of lampalizumab administered by intravitreal injections for approximately 96 weeks.
  Interventions: Drug: Lampalizumab
- Sham Comparator (Sham Comparator): Participants will receive sham comparator Q4W or Q6W for 96 weeks.
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Lampalizumab — Participants will receive 10 mg dose of lampalizumab administered intravitreally.
  Other Names: RO5490249
  Arms: Lampalizumab Once in Every 4 Weeks (Q4W); Lampalizumab Once in Every 6 Weeks (Q6W)
Other: Sham — A sham injection is a procedure that mimics an intravitreal injection of lampalizumab.
  Arms: Sham Comparator

SUMMARY:
This study is a Phase III, double-masked, multicenter, randomized, sham injection-controlled study evaluating the efficacy and safety of lampalizumab administered by intravitreal injections in participants with geographic atrophy (GA) secondary to age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Well demarcated area(s) of Geographic Atrophy (GA) secondary to Age-Related Macular Degeneration (AMD) with no evidence of prior or active choroidal neovascularization (CNV) in both eyes

Exclusion Criteria:

Ocular Exclusion Criteria: Study Eye

* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD
* Previous laser photocoagulation for CNV, diabetic macular edema, retinal vein occlusion, and proliferative diabetic retinopathy
* Previous intravitreal drug delivery (intravitreal corticosteroid injection, anti-angiogenic drugs, anti-complement agents, or device implantation) Ocular Exclusion Criteria: Both Eyes
* GA in either eye due to causes other than AMD
* Previous treatment with eculizumab, lampalizumab and/or fenretinide

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 906 (Actual)
Dates: Start 2014-09-18 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (145):
- United States (76):
  - Uni of Alabama At Birmingham Clinical Research Unit, Birmingham, Alabama
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retina Centers P.C., Tucson, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - The Gavin Herbert Eye Institute - UC, Irvine, Irvine, California
  - Jules Stein Eye Institute/ UCLA, Los Angeles, California
  - East Bay Retina Consultants, Oakland, California
  - Southern CA Desert Retina Cons, Palm Desert, California
  - W Coast Retina Med Group Inc, San Francisco, California
  - UCSF; Ophthalmology, San Francisco, California
  - Orange County Retina Med Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Florida Eye Microsurgical Inst, Boynton Beach, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Bascom Palmer Eye Institute, Palm Beach Gardens, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southern Vitreoretinal Assoc, Tallahassee, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - Northwestern Medical Group/Northwestern University, Chicago, Illinois
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Midwest Eye Institute Northside, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates, Shawnee Mission, Kansas
  - Lahey Clinic Med Ctr, Lexington, Kentucky
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Maine Eye Center, Portland, Maine
  - Retina Specialists, Towson, Maryland
  - Tufts Medical Center Research, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Vitreo-Retinal Associates, PC, Worcester, Massachusetts
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Specialty Eye Institute, Jackson, Michigan
  - Assoc Retinal Consultants PC, Royal Oak, Michigan
  - Retina Consultants of Michigan, Southfield, Michigan
  - Eye Surgical Associates, Lincoln, Nebraska
  - Retina Consultants of Nevada, Las Vegas, Nevada
  - Retina Center of New Jersey, Bloomfield, New Jersey
  - New Jersey Retina Research Foundation, Edison, New Jersey
  - Delaware Valley Retina Assoc, Lawrenceville, New Jersey
  - Long Is. Vitreoretinal Consult, Hauppauge, New York
  - Opthalmic Consultants of LI, Lynbrook, New York
  - New York Eye & Ear Infirmary, New York, New York
  - Retina Consultants of Western New York, Orchard Park, New York
  - Retina Vit Surgeons/Central NY, Syracuse, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Wake Forest Baptist Health Eye Centre, Winston-Salem, North Carolina
  - Retina Assoc of Cleveland Inc, Beachwood, Ohio
  - Cleveland Clinic Foundation; Cole Eye Institute, Cleveland, Ohio
  - Retina Vitreous Consultants, Monroeville, Pennsylvania
  - Associates in Ophthalmology, West Mifflin, Pennsylvania
  - Charleston Neuroscience Inst, Ladson, South Carolina
  - Tennessee Retina PC., Nashville, Tennessee
  - Vanderbilt, Nashville, Tennessee
  - Retina Res Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - UT Southwestern MC at Dallas, Dallas, Texas
  - Valley Retina Institute P.A., McAllen, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Eye Surgeons of Richmond Inc. dba Virginia Eye Institute, Richmond, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
  - Virginia Retina Center, Warrenton, Virginia
  - Retina Center Northwest, Silverdale, Washington
  - Spokane Eye Clinical Research, Spokane, Washington
  - West Virginia University Eye Institute, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
- Argentina (5):
  - Organizacion Medica de Investigacion, Buenos Aires
  - Fundacion Zambrano, CABA
  - Oftar, Mendoza
  - Microcirugía Ocular S.A, Rosario
  - Grupo Laser Vision, Rosario
- Australia (4):
  - Eyeclinic Albury Wodonga, Albury, New South Wales
  - Marsden Eye Research Centre, Parramatta, New South Wales
  - Save Sight Institute, Sydney, New South Wales
  - Sydney West Retina, Westmead, New South Wales
- Kepler Universitätskliniken GmbH - Med Campus III; Abt. für Augenheilkunde, Linz, Austria
- Belgium (4):
  - CHU Brugmann (Victor Horta), Brussels
  - UZ Gent, Ghent
  - UZ Leuven Sint Rafael, Leuven
  - CHU Sart-Tilman, Liège
- Canada (8):
  - Calgary Retina Consultants, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - QEII - HSC Department of Ophthalmology, Halifax, Nova Scotia
  - University of Ottawa Eye Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael'S Hospital, Toronto, Ontario
  - University Health Network Toronto Western Hospital, Toronto, Ontario
  - Institut De L'Oeil Des Laurentides, Boisbriand, Quebec
- Sjællands Universitetshospital, Roskilde; Øjenafdelingen, Roskilde, Denmark
- France (6):
  - Chi De Creteil; Ophtalmologie, Créteil
  - Centre Odeon; Exploration Ophtalmologique, Paris
  - Hopital Lariboisiere; Ophtalmologie, Paris
  - Centre Ophtalmologique; Imagerie et laser, Paris
  - Ch Pitie Salpetriere; Ophtalmologie, Paris
  - CHU Poitiers - CHR La Miletrie; Ophtalmologie, Poitiers
- Germany (7):
  - Universitäts-Augenklinik Bonn, Bonn
  - Universitätsklinikum Köln; Augenklinik, Cologne
  - Universitätsmedizin Göttingen Georg-August-Universität; Klinik für Augenheilkunde, Göttingen
  - Medizinische Hochschule Hannover, Klinik für Augenheilkunde, Hanover
  - Universitätskliniikum Schleswig-Holstein, Campus Lübeck, Klinik für Augenheilkunde, Lübeck
  - Augenabteilung am St. Franziskus-Hospital, Münster
  - Universitätsklinikum Münster; Augenheilkunde, Münster
- Hungary (3):
  - Budapest Retina Associates Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont; Szemeszeti Klinika, Debrecem
  - Ganglion Medial Center, Pécs
- Italy (4):
  - Fondazione Ptv Policlinico Tor Vergata Di Roma;U.O.S.D. Patologie Renitiche, Rome, Lazio
  - Fondazione G.B. Bietti Per Lo Studio E La Ricerca in Oftalmologia-Presidio Ospedaliero Britannico, Rome, Lazio
  - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico-Clinica Regina Elena;U.O.C Oculistica, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Di Sassari;U.O. Oculistica, Sassari, Sardinia
- Mexico (2):
  - Macula Retina Consultores, Mexico City
  - Hospital de la Ceguera APEC, Mexico City
- Netherlands (3):
  - Academisch Medisch Centrum Universiteit Amsterdam, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden
  - Radboud University Nijmegen Medical Centre; Ophthalmology, Nijmegen
- Peru (2):
  - CLINICA RICARDO PALMA; Oftalmologos Contreras, Lima
  - Clinica Anglo Americana, Lima
- Poland (4):
  - OFTALMIKA Sp. z o.o, Bydgoszcz
  - Optimum Profesorskie Centrum Okulistyki, Gdansk
  - Gabinet Okulistyczny Prof Edward Wylegala, Katowice
  - SP ZOZ Szpital Uniwersytecki w Krakowie Oddział Kliniczny Okulistyki i Onkologii Okulistycznej, Krakow
- Slovakia (3):
  - Nemocnica sv. Michala, a.s., Bratislava
  - Fakultna nemocnica Trencin Ocna klinika, Trenčín
  - Fakultna nemocnica s poliklinikou Zilina; Ocne oddelenie, Žilina
- Spain (7):
  - Hospital Universitari de Bellvitge; Servicio de Oftalmologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Catalunya, San Cugat Del Valles, Barcelona
  - Instituto Clinico Quirurgico de Oftalmologia - ICQO, Bilbao, Guipuzcoa
  - VISSUM Instituto Oftalmológico de Alicante, Alicante
  - Institut de la Macula i la retina, Barcelona
  - FISABIO. Fundación Oftalmologica del Mediterraneo, Valencia
  - Hospital Universitario Rio Hortega; Servicio de Oftalmologia, Valladolid
- Stadtspital Triemli; Augenklinik, Zurich, Switzerland
- United Kingdom (4):
  - Ayr Hospital, Ayr
  - The Princess Alexandra Eye Pavilion, Edinburgh
  - Frimley Park Hospital, Frimley
  - Royal Hallamshire Hospita, Sheffield

REFERENCES:
- [Derived] Salvi A, Cluceru J, Gao SS, Rabe C, Schiffman C, Yang Q, Lee AY, Keane PA, Sadda SR, Holz FG, Ferrara D, Anegondi N. Deep Learning to Predict the Future Growth of Geographic Atrophy from Fundus Autofluorescence. Ophthalmol Sci. 2024 Oct 23;5(2):100635. doi: 10.1016/j.xops.2024.100635. eCollection 2025 Mar-Apr. PMID 39758130
- [Derived] Cluceru J, Anegondi N, Gao SS, Lee AY, Lad EM, Chakravarthy U, Yang Q, Steffen V, Friesenhahn M, Rabe C, Ferrara D. Topographic Clinical Insights From Deep Learning-Based Geographic Atrophy Progression Prediction. Transl Vis Sci Technol. 2024 Aug 1;13(8):6. doi: 10.1167/tvst.13.8.6. PMID 39102242
- [Derived] Bressler NM, Freund KB, Bakri SJ, Kim JE, Ferrara D, Brittain C, Pickthorn K, Lin H, Sun C, Martin J. Intraocular Pressure Outcomes After Lampalizumab Injections in Patients With Geographic Atrophy. JAMA Ophthalmol. 2024 Aug 1;142(8):772-776. doi: 10.1001/jamaophthalmol.2024.2061. PMID 38900484
- [Derived] Chang DS, Callaway NF, Steffen V, Csaky K, Guymer RH, Birch DG, Patel PJ, Ip M, Gao SS, Briggs J, Honigberg L, Lai P, Ferrara D, Sepah YJ. Macular Sensitivity Endpoints in Geographic Atrophy: Exploratory Analysis of Chroma and Spectri Clinical Trials. Ophthalmol Sci. 2023 Jun 12;4(1):100351. doi: 10.1016/j.xops.2023.100351. eCollection 2024 Jan-Feb. PMID 37869030
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061
- [Derived] Miere A, Capuano V, Kessler A, Zambrowski O, Jung C, Colantuono D, Pallone C, Semoun O, Petit E, Souied E. Deep learning-based classification of retinal atrophy using fundus autofluorescence imaging. Comput Biol Med. 2021 Mar;130:104198. doi: 10.1016/j.compbiomed.2020.104198. Epub 2020 Dec 28. PMID 33383315
- [Derived] Heier JS, Pieramici D, Chakravarthy U, Patel SS, Gupta S, Lotery A, Lad EM, Silverman D, Henry EC, Anderesi M, Tschosik EA, Gray S, Ferrara D, Guymer R; Chroma and Spectri Study Investigators. Visual Function Decline Resulting from Geographic Atrophy: Results from the Chroma and Spectri Phase 3 Trials. Ophthalmol Retina. 2020 Jul;4(7):673-688. doi: 10.1016/j.oret.2020.01.019. Epub 2020 Jan 31. PMID 32199866
- [Derived] Holz FG, Sadda SR, Busbee B, Chew EY, Mitchell P, Tufail A, Brittain C, Ferrara D, Gray S, Honigberg L, Martin J, Tong B, Ehrlich JS, Bressler NM; Chroma and Spectri Study Investigators. Efficacy and Safety of Lampalizumab for Geographic Atrophy Due to Age-Related Macular Degeneration: Chroma and Spectri Phase 3 Randomized Clinical Trials. JAMA Ophthalmol. 2018 Jun 1;136(6):666-677. doi: 10.1001/jamaophthalmol.2018.1544. PMID 29801123

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 906 participants were randomized to the study from 131 investigation sites across 19 countries. The study was terminated early by the Sponsor due to lack of efficacy.
Pre-assignment Details: This study enrolled participants with bilateral Geographic Atrophy (GA) secondary to Age-Related Macular Degeneration (AMD) and no signs of prior or active choroidal neovascularization (CNV), age >= 50 years with a valid complement factor I (CFI)-profile biomarker result.
Groups:
- Sham Comparator: Participants received sham comparator once in every 4 weeks (Q4W) or once in every 6 weeks (Q6W) starting at Day 1 visit.
- Lampalizumab Q4W: Participants received 10 milligrams (mg) dose of lampalizumab administered by intravitreal injections Q4W starting at Day 1 visit.
- Lampalizumab Q6W: Participants received 10 mg dose of lampalizumab administered by intravitreal injections Q6W starting at Day 1 visit.
Period: Overall Study
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Started | 305 | 298 | 303
Completed | 163 | 160 | 165
Not Completed | 142 | 138 | 138
Not completed — Adverse Event | 8 | 9 | 8
Not completed — Death | 5 | 4 | 6
Not completed — Lost to Follow-up | 3 | 3 | 1
Not completed — Non-compliance | 0 | 0 | 1
Not completed — Withdrawal by Subject | 25 | 29 | 24
Not completed — Study Terminated by Sponsor | 98 | 88 | 94
Not completed — Physician Decision | 1 | 0 | 2
Not completed — Unspecified Reason | 2 | 5 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all the participants who were randomized to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W | Total
Number analyzed (Participants) | 305 | 298 | 303 | 906
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.5 (7.8) | 77.5 (7.9) | 78.3 (8.5) | 78.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 182 | 185 | 553
  Male | 119 | 116 | 118 | 353
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 1
  White | 302 | 294 | 295 | 891
  Multiple | 0 | 0 | 1 | 1
  Unknown | 3 | 2 | 6 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 17 | 18 | 55
  Not Hispanic or Latino | 279 | 278 | 282 | 839
  Not Stated | 2 | 3 | 1 | 6
  Unknown | 4 | 0 | 2 | 6
Geographic Atrophy (GA) Area, as Assessed by Fundus Autofluoresence (FAF) [Mean (Standard Deviation); unit: millimeter square (mm^2)] — At baseline the area of GA was assessed by FAF. Population: ITT population included all the participants who were randomized to the study. Reported here are the number of participants for whom data was collected.
  millimeter square (mm^2)
    number analyzed (Participants) | 305 | 298 | 302 | 905
    (all) | 7.953 (3.925) | 7.910 (3.887) | 8.116 (4.236) | 7.993 (4.016)
Number of Absolute Scotomatous Points as Assessed by Mesopic Micrometry [Mean (Standard Deviation); unit: absolute scotomatous points] — Scotomatous points were the testing points on microperimetry examination that were centered on the macula and reported a lack of retinal sensitivity within the range tested, a maximum of 68 points were tested within this range. Higher results indicate expansion of absolute scotoma and higher number of abolute scotomatous points. Mesopic microperimetry assessments were performed post-dilation on the study eye only, and the data was forwarded to the central reading center. Population: The microperimetry analysis population consisted of all participants who met the microperimetry eligibility criteria assessed by the reading center (participants at selected sites only; participants grouped according to treatment assigned at randomization).
  absolute scotomatous points
    number analyzed (Participants) | 44 | 33 | 39 | 116
    (all) | 29.1 (16.8) | 25.2 (13.4) | 20.5 (13.4) | 25.1 (15.1)
Macular Sensitivity as Assessed by Mesopic Microperimetry [Mean (Standard Deviation); unit: decibel (dB)] — Mesopic microperimetry was used to assess macular sensitivity and assessments were performed post-dilation on the study eye only, and the data was forwarded to the central reading center. Population: The microperimetry analysis population consisted of all participants who met the microperimetry eligibility criteria assessed by the reading center (participants at selected sites only; participants grouped according to treatment assigned at randomization).
  decibel (dB)
    number analyzed (Participants) | 44 | 33 | 39 | 116
    (all) | 5.40 (3.37) | 6.37 (4.02) | 7.38 (3.40) | 6.34 (3.64)
Best Corrected Visual Acuity (BCVA) Score as Assessed by Early Treatment Diabetic Retinopathy Study [Mean (Standard Deviation); unit: letters] — BCVA score was based on the number of letters read correctly on the ETDRS visual acuity chart assessed at a starting distance of 4 meters. BCVA score testing was performed prior to dilating the eyes. BCVA score ranges from 0 to 100 letters in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). Population: ITT population included all the participants who were randomized to the study. Reported here are the number of participants for whom data was collected.
  letters
    number analyzed (Participants) | 301 | 295 | 301 | 897
    (all) | 65.9 (9.9) | 66.1 (10.0) | 66.4 (10.1) | 66.2 (10.0)
Low Luminance Visual Acuity (LLVA) as Assessed by ETDRS Chart Under Low Luminance Conditions [Mean (Standard Deviation); unit: letters] — The LLVA was measured by placing a 2.0-log-unit neutral density filter over the best correction for that eye and having the participant read the normally illuminated ETDRS chart. The assessment was performed prior to dilating the eyes. LLVA score ranges from 0 to 100 letters in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). Population: ITT population included all the participants who were randomized to the study. Reported here are the number of participants for whom data was collected.
  letters
    number analyzed (Participants) | 299 | 287 | 293 | 879
    (all) | 36.0 (15.7) | 36.9 (17.8) | 36.2 (16.7) | 36.4 (16.7)
Binocular Reading Speed as Assessed by Minnesota Low-Vision Reading Test or Radner Reading Charts [Mean (Standard Deviation); unit: words per minute (wpm)] — Minnesota Low-Vision Reading (MNRead) acuity cards were continuous-text reading-acuity cards suitable for measuring reading acuity and reading speed of normal and low-vision participants. A stopwatch was used to record time to a tenth of a second. Sentences that could not be read or were not attempted due to vision should be recorded as 0 for time and 10 for errors. Radner Reading Cards were suitable for measuring reading speed, reading visual acuity, and critical print size. Reading test was stopped when reading time was longer than 20 seconds or when participant was making severe errors. Population: ITT population included all the participants who were randomized to the study. Reported here are the number of participants for whom data was collected.
  words per minute (wpm)
    number analyzed (Participants) | 278 | 262 | 269 | 809
    (all) | 106.89 (57.98) | 109.18 (60.14) | 104.22 (62.37) | 106.74 (60.12)
National Eye Institute Visual Functioning Questionnaire 25-item (NEI VFQ-25) Version Composite Score [Mean (Standard Deviation); unit: score on a scale] — NEI-VFQ-25 questionnaire included 25 items based on which overall composite VFQ score and 12 subscales were derived: near activities, distance activities, general health,general vision, ocular pain, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision and peripheral vision. Response to each question converted to 0-100 score. Each subscale, total score=average of items contributing to score. For each subscale and total score, score range: 0 to 100, a higher score represents better functioning. Population: ITT population included all the participants who were randomized to the study. Reported here are the number of participants for whom data was collected.
  score on a scale
    number analyzed (Participants) | 276 | 275 | 282 | 833
    (all) | 66.16 (17.33) | 64.80 (16.12) | 65.19 (17.27) | 65.38 (16.91)
Mean Functional Reading Independence (FRI) Index [Mean (Standard Deviation); unit: score on a scale] — The FRI was an interviewer-administered questionnaire with 7-items on functional reading activities most relevant to GA AMD participants. It has one total index score. For each FRI Index reading activity performed in the past 7 days, participants were asked about the extent to which they required vision aids, adjustments in the activity, or help from another participant. Mean FRI Index scores range from 1 to 4, with higher scores indicating greater independence. Population: ITT population included all the participants who were randomized to the study. Reported here are the number of participants for whom data was collected.
  score on a scale
    number analyzed (Participants) | 276 | 273 | 280 | 829
    (all) | 2.69 (0.83) | 2.71 (0.79) | 2.70 (0.82) | 2.70 (0.81)
NEI VFQ-25 Near Activity Subscale Score [Mean (Standard Deviation); unit: score on a scale] — NEI-VFQ-25 questionnaire included 25 items based on near activities, which are defined as reading ordinary print in newspapers, performing work or hobbies requiring near vision, or finding something on a crowded shelf. Response to each question converted to 0-100 score. Subscale=average of items contributing to score. For this subscale the score range is 0 to 100, a higher score represents better functioning. Population: ITT population included all the participants who were randomized to the study. Reported here are the number of participants for whom data was collected.
  score on a scale
    number analyzed (Participants) | 276 | 275 | 282 | 833
    (all) | 54.98 (20.98) | 53.78 (20.56) | 53.67 (22.21) | 54.14 (21.25)
NEI VFQ-25 Distance Activity Subscale Score [Mean (Standard Deviation); unit: score on a scale] — NEI-VFQ-25 questionnaire included 25 items based on which distance activities was measured. Distance activities are defined as reading street signs or names on stores, and going down stairs, steps, or curbs. Response to each question converted to 0-100 score. Subscale=average of items contributing to score. For this subscale the score range is 0 to 100, a higher score represents better functioning. Population: ITT population included all the participants who were randomized to the study. Reported here are the number of participants for whom data was collected.
  score on a scale
    number analyzed (Participants) | 276 | 275 | 282 | 833
    (all) | 62.86 (21.46) | 60.97 (20.48) | 62.10 (22.16) | 61.98 (21.37)
Monocular Maximum Reading Speed as Assessed by MNRead Charts or Radner Reading Charts [Mean (Standard Deviation); unit: wpm] — MNRead acuity cards were continuous-text reading-acuity cards suitable for measuring the reading acuity and reading speed of normal and low-vision participants. A stopwatch was used to record time to a tenth of a second. Sentences that could not be read or were not attempted due to vision should be recorded as 0 for time and 10 for errors. Radner Reading Cards were suitable for measuring reading speed, reading visual acuity, and critical print size. Reading test was stopped when reading time was longer than 20 seconds or when participant was making severe errors. Population: ITT population included all the participants who were randomized to the study. Reported here are the number of participants for whom data was collected.
  wpm
    number analyzed (Participants) | 278 | 265 | 271 | 814
    (all) | 80.89 (52.95) | 85.18 (54.55) | 79.49 (54.23) | 81.82 (53.89)
GA Area in Complement Factor I (CFI) Positive Participants [Mean (Standard Deviation); unit: mm^2] — For CFI profile, positive biomarker status refers to the presence (carrier) of the risk allele at CFI and at least one risk allele at complement factor H (CFH) or risk locus containing both complement component 2 and complement factor B (C2/CFB). Population: ITT population included all the participants who were randomized to the study. Reported here are the number of participants for whom data was collected.
  mm^2
    number analyzed (Participants) | 181 | 176 | 177 | 534
    (all) | 8.015 (3.915) | 8.152 (4.118) | 8.406 (4.399) | 8.190 (4.142)
GA Area in CFI Negative Participants [Mean (Standard Deviation); unit: mm^2] — For CFI profile, negative biomarker status refers to the absence of the risk allele at CFI and at least one risk allele at CFH or C2/CFB. Population: ITT population included all the participants who were randomized to the study. Reported here are the number of participants for whom data was collected.
  mm^2
    number analyzed (Participants) | 124 | 122 | 125 | 371
    (all) | 7.864 (3.952) | 7.560 (3.515) | 7.705 (3.975) | 7.710 (3.814)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Geographic Atrophy (GA) Area, as Assessed by Fundus Autofluoresence (FAF) at Week 48
Description: The change in GA lesion area was measured by FAF and analysis of FAF images was performed by the central reading center. A positive change from baseline indicates an increase in size of GA lesion area (worsening; disease progression).
Time Frame: Baseline, Week 48
Population: ITT population included all the participants who were randomized to the study. Participants analyzed in this outcome measure were those included in Mixed-effect model repeated measures (MMRM) analysis.
Measure: Mean (Standard Error); unit: millimeter square (mm^2)
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 274 | 259 | 270
millimeter square (mm^2) | 2.035 (0.066) | 2.016 (0.068) | 2.086 (0.067)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, visit, treatment-by-visit interaction, baseline GA area, lesion location, contiguity, biomarker status, modified baseline BCVA and sex; Test type: Superiority; p = 0.8381, MMRM; Difference in Adjusted Means = -0.019, 95% CI 2-sided [-0.206 to 0.167]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5901, MMRM; Difference in Adjusted Means = 0.051, 95% CI 2-sided [-0.134 to 0.236]

2. Secondary Outcome: Change From Baseline in Number of Absolute Scotomatous Points as Assessed by Mesopic Micrometry at Week 48
Description: Scotomatous points were the testing points on microperimetry examination that were centered on the macula and reported a lack of retinal sensitivity within the range tested, a maximum of 68 points were tested within this range. Higher results indicate expansion of absolute scotoma and higher number of abolute scotomatous points. Mesopic microperimetry assessments were performed post-dilation on the study eye only, and the data was forwarded to the central reading center. The data was collected up to Week 48 instead of Week 96, due to early termination of the study. A positive change from baseline indicates an increase in the number of absolute scotomatous points (more lack of retinal sensitivity); disease worsening.
Time Frame: Baseline, Week 48
Population: The microperimetry analysis population consisted of all participants who met the microperimetry eligibility criteria assessed by the reading center (participants at selected sites only; participants grouped according to treatment assigned at randomization). Participants analyzed in this outcome measure were those included in MMRM analysis.
Measure: Mean (Standard Error); unit: absolute scotomatous points
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 30 | 26 | 26
absolute scotomatous points | 8.3 (1.7) | 8.1 (1.8) | 8.3 (1.8)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, visit, treatment-by-visit interaction, baseline number of absolute scotomatous points, GA lesion location, contiguity, biomarker status, modified baseline BCVA and sex; Test type: Superiority; p = 0.9350, MMRM; Difference in Adjusted Means = -0.2, 95% CI 2-sided [-5.2 to 4.8]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.9789, MMRM; Difference in Adjusted Means = 0.1, 95% CI 2-sided [-5.0 to 5.2]

3. Secondary Outcome: Change From Baseline in Mean Macular Sensitivity as Assessed by Mesopic Microperimetry at Week 48
Description: Mesopic microperimetry was used to assess macular sensitivity and assessments were performed post-dilation on the study eye only, and the data was forwarded to the central reading center. A negative change from baseline indicates a decrease in the mean macular sensitivity; disease worsening. The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 2
Measure: Mean (Standard Error); unit: decibel (dB)
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 30 | 26 | 26
decibel (dB) | -1.61 (0.33) | -1.33 (0.34) | -2.24 (0.35)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, visit, treatment-by-visit interaction, baseline mean macular sensitivity, GA lesion location, contiguity, biomarker status, modified baseline BCVA and sex; Test type: Superiority; p = 0.5538, MMRM; Difference in Adjusted Means = 0.28, 95% CI 2-sided [-0.66 to 1.22]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.2032, MMRM; Difference in Adjusted Means = -0.63, 95% CI 2-sided [-1.60 to 0.35]

4. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Score as Assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) Chart at Week 48
Description: BCVA score was based on the number of letters read correctly on the ETDRS visual acuity chart assessed at a starting distance of 4 meters (m). BCVA score testing was performed prior to dilating the eyes. BCVA score ranges from 0 to 100 letters in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A negative change from baseline indicates a decrease in the visual acuity; disease worsening. The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: ITT population included all the participants who were randomized to the study. Participants analyzed in this outcome measure were those included in MMRM analysis.
Measure: Mean (Standard Error); unit: letters
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 267 | 259 | 261
letters | -4.5 (0.6) | -3.4 (0.6) | -4.6 (0.6)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, visit, treatment-by-visit interaction, baseline BCVA, GA lesion location, biomarker status, and sex; Test type: Superiority; p = 0.2547, MMRM; Difference in Adjusted Means = 1.0, 95% CI 2-sided [-0.7 to 2.8]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.8423, MMRM; Difference in Adjusted Means = -0.2, 95% CI 2-sided [-1.9 to 1.6]

5. Secondary Outcome: Percentage of Participants With Less Than 15 Letters Loss From Baseline in BCVA Score at Week 48
Description: Loss of less than 15 letters from baseline was assessed by the ETDRS chart at a starting distance of 4 meters (m). BCVA was measured using an eye chart and was reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Week 48
Population: ITT population included all the participants who were randomized to the study. Reported here is the number of participants for whom data were collected.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 267 | 259 | 262
percentage of participants | 85.8 [81.6 to 90.0] | 88.8 [85.0 to 92.6] | 87.0 [83.0 to 91.1]
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: The adjusted analysis was based on a logistic regression analysis. The model included terms for treatment group, baseline BCVA, baseline GA lesion location, biomarker status, and sex; Test type: Superiority; p = 0.3248, Regression, Logistic; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.8 to 2.2]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.7209, Regression, Logistic; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.7 to 1.8]

6. Secondary Outcome: Change From Baseline in Low Luminance Visual Acuity (LLVA) as Assessed by ETDRS Chart Under Low Luminance Conditions at Week 48
Description: The LLVA was measured by placing a 2.0-log-unit neutral density filter over the best correction for that eye and having the participant read the normally illuminated ETDRS chart. The assessment was performed prior to dilating the eyes. LLVA score ranges from 0 to 100 letters in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: letters
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 265 | 251 | 252
letters | -3.0 (0.7) | -2.4 (0.7) | -2.7 (0.7)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, visit, treatment-by-visit interaction, baseline LLVA, GA lesion location, biomarker status, modified baseline BCVA ETDRS chart Snellen equivalent category, and sex; Test type: Superiority; p = 0.5695, MMRM; Difference in Adjusted Means = 0.6, 95% CI 2-sided [-1.4 to 2.6]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.7865, MMRM; Difference in Adjusted Means = 0.3, 95% CI 2-sided [-1.7 to 2.3]

7. Secondary Outcome: Percentage of Participants With Less Than 15 Letters Loss From Baseline in LLVA Score at Week 48
Description: Loss of less than 15 letters from baseline was assessed by the ETDRS chart at a starting distance of 4 m. The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Week 48
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 265 | 251 | 253
percentage of participants | 86.8 [82.7 to 90.9] | 85.3 [80.9 to 89.6] | 86.6 [82.4 to 90.8]
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: The adjusted analysis was based on a logistic regression analysis. The model included terms for treatment group, baseline LLVA, baseline GA lesion location, biomarker status, modified baseline BCVA ETDRS chart Snellen equivalent category, and sex; Test type: Superiority; p = 0.9448, Regression, Logistic; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.6 to 1.7]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.8764, Regression, Logistic; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.6 to 1.8]

8. Secondary Outcome: Change From Baseline in Binocular Reading Speed as Assessed by Minnesota Low-Vision Reading Test (MNRead) Charts or Radner Reading Charts at Week 48
Description: MNRead acuity cards were continuous-text reading-acuity cards suitable for measuring the reading acuity and reading speed of normal and low-vision participants. The MNRead acuity cards consisted of single, simple sentences with equal numbers of characters. A stopwatch was used to record time to a tenth of a second. Sentences that could not be read or were not attempted due to vision should be recorded as 0 for time and 10 for errors. The Radner Reading Cards were suitable for measuring reading speed, reading visual acuity, and critical print size. The reading test was stopped when the reading time was longer than 20 seconds or when the participant was making severe errors. A negative change from baseline indicates a decrease in the binocular reading speed; disease worsening. The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: words per minute (wpm)
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 242 | 223 | 229
words per minute (wpm) | -18.97 (2.37) | -13.32 (2.47) | -19.96 (2.44)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, baseline maximum reading speed, type of reading charts, baseline BCVA of better seeing eye, biomarker status, and sex; Test type: Superiority; p = 0.0991, MMRM; Difference in Adjusted Means = 5.66, 95% CI 2-sided [-1.07 to 12.38]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.7713, MMRM; Difference in Adjusted Means = -0.99, 95% CI 2-sided [-7.66 to 5.69]

9. Secondary Outcome: Change From Baseline in Monocular Maximum Reading Speed as Assessed by MNRead Charts or Radner Reading Charts at Week 48
Description: MNRead acuity cards were continuous-text reading-acuity cards suitable for measuring the reading acuity and reading speed of normal and low-vision participants. The MNRead acuity cards consisted of single, simple sentences with equal numbers of characters. A stopwatch was used to record time to a tenth of a second. Sentences that could not be read or were not attempted due to vision should be recorded as 0 for time and 10 for errors. The Radner Reading Cards were suitable for measuring reading speed, reading visual acuity, and critical print size. The reading test was stopped when the reading time was longer than 20 seconds or when the participant was making severe errors. A negative change from baseline indicates a decrease in the monocular reading speed; disease worsening. The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: wpm
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 243 | 229 | 233
wpm | -19.63 (2.41) | -17.91 (2.49) | -18.16 (2.47)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; MMRM analysis uses change as response variable included terms for treatment group, baseline maximum reading speed, type of reading charts, biomarker status, modified baseline BCVA and sex; Test type: Superiority; p = 0.6204, MMRM; Difference in Adjusted Means = 1.72, 95% CI 2-sided [-5.09 to 8.53]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.6705, MMRM; Difference in Adjusted Means = 1.47, 95% CI 2-sided [-5.31 to 8.25]

10. Secondary Outcome: Change From Baseline in National Eye Institute Visual Functioning Questionnaire 25-item (NEI VFQ-25) Version Composite Score at Week 48
Description: NEI-VFQ-25 questionnaire included 25 items based on which overall composite VFQ score and 12 subscales were derived: near activities, distance activities, general health,general vision, ocular pain, vision-specific social functioning, vision-specific mental health, vision-specific role difficulties, vision-specific dependency, driving, color vision and peripheral vision. Response to each question converted to 0-100 score. Each subscale, total score=average of items contributing to score. For each subscale and total score, score range: 0 to 100, a higher score represents better functioning. A negative change from baseline indicates a decrease in the visual functioning; disease worsening. The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 239 | 234 | 248
scores on a scale | -1.31 (0.71) | -1.66 (0.72) | -2.87 (0.70)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q6W; Week 48: MMRM analysis uses change as response variable and included treatment group, baseline score, baseline BCVA of better seeing eye, biomarker status, and sex; Test type: Superiority; p = 0.7246, MMRM; Difference in Adjusted Means = -0.36, 95% CI 2-sided [-2.35 to 1.64]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.1193, MMRM; Difference in Adjusted Means = -1.56, 95% CI 2-sided [-3.53 to 0.40]

11. Secondary Outcome: Change From Baseline in NEI VFQ-25 Near Activity Subscale Score at Week 48
Description: NEI-VFQ-25 questionnaire included 25 items based on which near activities were measured. Near activities are defined as reading ordinary print in newspapers, performing work or hobbies requiring near vision, or finding something on a crowded shelf. Response to each question converted to 0-100 score. Subscale=average of items contributing to score. For this subscale the score range is 0 to 100, a higher score represents better functioning. A negative change from baseline indicates a decrease in the near visual activities; disease worsening. The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 239 | 234 | 248
score on a scale | -2.12 (0.93) | -2.35 (0.94) | -4.06 (0.92)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.8659, MMRM; Difference in Adjusted Means = -0.22, 95% CI 2-sided [-2.84 to 2.39]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.1399, MMRM; Difference in Adjusted Means = -1.94, 95% CI 2-sided [-4.51 to 0.64]

12. Secondary Outcome: Change From Baseline in NEI VFQ-25 Distance Activity Subscale Score at Week 48
Description: NEI-VFQ-25 questionnaire included 25 items based on which distance activities were measured. Distance activities are defined as reading street signs or names on stores, and going down stairs, steps, or curbs. Response to each question converted to 0-100 score. Subscale=average of items contributing to score. For this subscale the score range is 0 to 100, a higher score represents better functioning. A negative change from baseline indicates a decrease in the distance visual activities; disease worsening. The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 239 | 234 | 248
score on a scale | -2.03 (0.99) | -1.04 (1.00) | -3.62 (0.97)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.4855, MMRM; Difference in Adjusted Means = 0.99, 95% CI 2-sided [-1.79 to 3.76]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.2515, MMRM; Difference in Adjusted Means = -1.60, 95% CI 2-sided [-4.33 to 1.13]

13. Secondary Outcome: Change From Baseline in Mean Functional Reading Independence (FRI) Index at Week 48
Description: The FRI was an interviewer-administered questionnaire with 7 items on functional reading activities most relevant to GA AMD participants. It has one total index score. For each FRI Index reading activity performed in the past 7 days, participants were asked about the extent to which they required vision aids, adjustments in the activity, or help from another participant. Mean FRI Index scores range from 1 to 4, with higher scores indicating greater independence. A negative change from baseline indicates a decrease in the FRI; disease worsening. The data was collected up to Week 48 instead of Week 96, due to early termination of the study.
Time Frame: Baseline, Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 237 | 230 | 244
score on a scale | -0.06 (0.04) | -0.13 (0.04) | -0.15 (0.04)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; Week 48: MMRM analysis uses change as response variable and included treatment group, baseline Mean FRI Index score, baseline BCVA of better seeing eye, biomarker status, and sex; Test type: Superiority; p = 0.2075, MMRM; Difference in Adjusted Means = -0.07, 95% CI 2-sided [-0.18 to 0.04]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.1222, MMRM; Difference in Adjusted Means = -0.08, 95% CI 2-sided [-0.19 to 0.02]

14. Primary Outcome: Change From Baseline in GA Area in Complement Factor I (CFI) Positive and Negative Participants at Week 48
Description: For CFI profile, positive or negative biomarker status refers to the presence (carrier) or absence of the risk allele at CFI and at least one risk allele at complement factor H (CFH) or risk locus containing both complement component 2 and complement factor B (C2/CFB).The change in GA lesion area was measured by FAF and analysis of FAF images was performed by the central reading center. A positive change from baseline indicates an increase in size of GA lesion area (worsening; disease progression).
Time Frame: Baseline, Week 48
Population: ITT population included all the participants who were randomized to the study. The analysis was done specifically for CFI-positive and negative participants. Number analyzed for each row signifies the participants evaluated for specified categories for each reporting group.
Measure: Mean (Standard Error); unit: mm^2
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
Number analyzed (Participants) | 305 | 298 | 303
mm^2
  CFI-Positive Participants: number analyzed (Participants) | 162 | 152 | 160
  CFI-Positive Participants | 2.067 (0.086) | 2.045 (0.089) | 2.144 (0.087)
  CFI-Negative Participants: number analyzed (Participants) | 112 | 107 | 110
  CFI-Negative Participants | 2.006 (0.103) | 1.974 (0.105) | 2.012 (0.104)
Statistical Analysis 1: Comparison: Sham Comparator vs Lampalizumab Q4W; CFI Positive: MMRM analysis uses change as response variable and included treatment group, visit, treatment-by-visit interaction, baseline GA area, lesion location, contiguity, biomarker status, modified baseline BCVA and sex; Test type: Superiority; p = 0.8612, MMRM; Difference in Adjusted Means = -0.022, 95% CI 2-sided [-0.266 to 0.223]
Statistical Analysis 2: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.5317, MMRM; Difference in Adjusted Means = 0.077, 95% CI 2-sided [-0.165 to 0.319]
Statistical Analysis 3: Comparison: Sham Comparator vs Lampalizumab Q4W; CFI Negative: MMRM analysis uses change as response variable and included treatment group, visit, treatment-by-visit interaction, baseline GA area, lesion location, contiguity, biomarker status, modified baseline BCVA and sex; Test type: Superiority; p = 0.8240, MMRM; Difference in Adjusted Means = -0.033, 95% CI 2-sided [-0.322 to 0.257]
Statistical Analysis 4: Comparison: Sham Comparator vs Lampalizumab Q6W; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p = 0.9676, MMRM; Difference in Adjusted Means = 0.006, 95% CI 2-sided [-0.283 to 0.294]

ADVERSE EVENTS:
Time Frame: Up to approximately 2 years
Description: Safety population included all participants who received at least one dose of study drug.
Arm/Group | Sham Comparator | Lampalizumab Q4W | Lampalizumab Q6W
All-Cause Mortality (participants affected / at risk) | 6/300 | 5/298 | 6/303
Serious Adverse Events (participants affected / at risk) | 97/300 | 118/298 | 108/303
Other Adverse Events (participants affected / at risk) | 221/300 | 239/298 | 232/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Comparator (N=300) | Lampalizumab Q4W (N=298) | Lampalizumab Q6W (N=303)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 3 | 3
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 4 | 3
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 0 | 2
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 3 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 3 | 6
Coronary artery disease (Cardiac disorders) | 4 | 1 | 2
Myocardial infarction (Cardiac disorders) | 0 | 1 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Diverticular hernia (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastric volvulus (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 2
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Chest pain (General disorders) | 1 | 1 | 2
Death (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 3 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1
Cystitis (Infections and infestations) | 1 | 0 | 2
Device related infection (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 2
Infection (Infections and infestations) | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 2 | 0
Perihepatic abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 9 | 11 | 5
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 3 | 3 | 2
Septic shock (Infections and infestations) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 3 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 2 | 4
Femur fracture (Injury, poisoning and procedural complications) | 1 | 4 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 3 | 3 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Internal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 2 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Blood pressure increased (Investigations) | 1 | 0 | 0
Heart rate irregular (Investigations) | 0 | 1 | 0
Myocardial necrosis marker increased (Investigations) | 0 | 1 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Benign neoplasm of ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Malignant melanoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 2
Cerebral microangiopathy (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 3 | 1
Cervicogenic vertigo (Nervous system disorders) | 1 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Dural arteriovenous fistula (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 2 | 0
Seizure (Nervous system disorders) | 1 | 0 | 1
Senile dementia (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 4 | 1
Vertigo CNS origin (Nervous system disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Bladder cyst (Renal and urinary disorders) | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 3 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 2 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
Blood pressure inadequately controlled (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 2 | 0
Hypotension (Vascular disorders) | 1 | 0 | 2
May-Thurner syndrome (Vascular disorders) | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 2 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Blindness transient (Eye disorders) | 0 | 2 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 1
Borderline glaucoma (Eye disorders) | 0 | 1 | 0
Choroidal neovascularisation (Eye disorders) | 2 | 2 | 1
Iritis (Eye disorders) | 0 | 1 | 1
Neovascular age-related macular degeneration (Eye disorders) | 3 | 3 | 3
Open angle glaucoma (Eye disorders) | 0 | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 2 | 0
Retinal neovascularisation (Eye disorders) | 0 | 0 | 1
Retinal tear (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 10 | 12 | 8
Visual acuity reduced transiently (Eye disorders) | 0 | 2 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1
Vitritis (Eye disorders) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Endophthalmitis (Infections and infestations) | 0 | 2 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyphaema (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 16 | 14
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Dry age-related macular degeneration (Eye disorders) | 2 | 0 | 2
Cataract (Eye disorders) | 0 | 0 | 1
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Comparator (N=300) | Lampalizumab Q4W (N=298) | Lampalizumab Q6W (N=303)
Conjunctival haemorrhage (Eye disorders) | 84 | 111 | 93
Eye pain (Eye disorders) | 20 | 39 | 33
Vitreous floaters (Eye disorders) | 16 | 41 | 25
Vitreous detachment (Eye disorders) | 24 | 22 | 24
Dry eye (Eye disorders) | 25 | 23 | 14
Cataract (Eye disorders) | 12 | 22 | 15
Posterior capsule opacification (Eye disorders) | 14 | 21 | 13
Intraocular pressure increased (Investigations) | 9 | 42 | 27
Nausea (Gastrointestinal disorders) | 15 | 10 | 7
Bronchitis (Infections and infestations) | 22 | 29 | 26
Fall (Injury, poisoning and procedural complications) | 36 | 29 | 34
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 20 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 21 | 15
Headache (Nervous system disorders) | 7 | 20 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 16 | 13
Hypertension (Vascular disorders) | 14 | 16 | 13
Urinary tract infection (Infections and infestations) | 25 | 26 | 21
Upper respiratory tract infection (Infections and infestations) | 17 | 14 | 11
Influenza (Infections and infestations) | 12 | 14 | 16
Retinal haemorrhage (Eye disorders) | 20 | 14 | 17
Punctate keratitis (Eye disorders) | 15 | 16 | 16
Nasopharyngitis (Infections and infestations) | 27 | 45 | 34

LIMITATIONS AND CAVEATS:
This study was terminated early by the Sponsor because the compound had demonstrated to lack of efficacy. Thus, not all participants in this study completed the full duration of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT02247479/SAP_000.pdf
  • Study Protocol (2015-09-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT02247479/Prot_001.pdf